CLINICAL TRIAL: NCT06465472
Title: Evaluation of the Efficacy and Safety of Stiripentol in Patients 6 Years and Older With Primary Hyperoxaluria Type 1, 2 or 3
Acronym: CRYSTAL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocodex (Industry)
Collaborators: Exystat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRYSTAL - STP226; 2023-508062-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-03; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Primary Hyperoxaluria Type 1; Primary Hyperoxaluria Type 2; Primary Hyperoxaluria Type 3
Keywords: Stiripentol; Primary Hyperoxaluria; Oxalate
MeSH Terms: conditions — Primary hyperoxaluria type 1; Primary hyperoxaluria type 2; Hyperoxaluria, Primary | interventions — stiripentol

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 periods: a 6-month, placebo-controlled, double-blind treatment period on which the primary endpoint will be evaluated (period 1) followed by a 6-month open-label treatment period with blind maintained on results (period 2).
  Patients who benefit from the treatment after the first 12 months of study treatment will be proposed to enter the 4 years open-label extension (OLE) part of the study to continue to assess the long-term efficacy and safety of stiripentol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All Sponsor personnel will be blinded to study drug treatment until the 6-month treatment period data is unblinded for the primary analysis. To ensure that blinding will be maintained along the study, the following measures are implemented:
  * the capsules are identical for both products
  * all packaging items, bottles (primary packagings) and boxes (secondary, tertiary and quaternary packagings) are identical bearing similar study specific labels.
  At the start of the open-label Period 2), in order to maintain the blind to treatment assignment, gradual initiation of treatment will be done in all patients over the first three days as follows: 30 mg/kg/day at Day1, 40 mg/kg/day at Day 2 and 50 mg/kg/day from Day 3 (with a maximum dose of 3,000 mg/day).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stiripentol (Experimental): Patients in this arms will receive 50 mg/kg/day oral stiripentol during the first 6 months double-blind placebo-controlled study period 1 (Day 1 through Month 6) then continue the same treatment for the following 6 months (period 2).
  Interventions: Drug: Stiripentol Oral Capsule; Biological: Urine samples collect; Biological: Blood samples collect; Other: Kidney imaging; Other: Quality of Life questionnaires
- Placebo (Placebo Comparator): Patients in this arms will receive 50 mg/kg/day oral placebo during the first 6 months double-blind placebo-controlled study period 1 (Day 1 through Month 6) then patients receiving placebo will switch over the 6 to 12 month-period to stiripentol (period 2).
  Interventions: Drug: Placebo Oral Capsule; Biological: Urine samples collect; Biological: Blood samples collect; Other: Kidney imaging; Other: Quality of Life questionnaires

INTERVENTIONS:
Drug: Stiripentol Oral Capsule — The target dose of stiripentol will be 50 mg/kg/day with a maximum dose of 3,000 mg/day. Patients allocated to the Stiripentol group will receive this treatment during the first 6 months, and in continuation up to 12 months.
  Arms: Stiripentol
Drug: Placebo Oral Capsule — Placebo capsules will be administered for the first 6 months. Then patients will switch to stiripentol over the 6- to 12-month period.
  Arms: Placebo
Biological: Urine samples collect — Collections of urine over 24 hours and the first urine in the morning (spot urines) will be carried out. Urine collections will be performed either during hospitalizations, or at home if appropriate conditions are met.
Biological: Blood samples collect — Series of blood samples will be taken (serum pregnancy test, Primary Hyperoxaluria genetic characterization, clinical laboratory assessments, vitamin B6 dosage, plasma oxalate dosage, stiripentol pharmacokinetics)
Other: Kidney imaging — Kidney imaging will be obtained. Renal ultrasounds will be compulsory for all patients.
Other: Quality of Life questionnaires — Kidney Disease Quality of Life Questionnaire : KDQOL-36 for patients ≥18 years of age at screening, and the Pediatric Quality of Life Inventory (PedsQL) including the generic and KF modules (parent and/or self-report versions) for patients <18 years of age at screening.
  EQ-5D: a standardized instrument consisting of a questionnaire and a visual analog scale pertaining to 5 dimensions. Scoring of the questionnaire is based on degrees of disability. Scoring of the visual analog scale is based on a visual scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicate better health status. The EQ-5D-5L questionnaire (will be utilized in patients ≥18 years of age at screening, and the EQ-5D-Y questionnaire will be utilized in patients <18 years of age at screening, where available.

SUMMARY:
Evaluation of the efficacy and safety of stiripentol in patients 6 years and older with primary hyperoxaluria type 1, 2 or 3.

DETAILED DESCRIPTION:
A multicenter randomized, double-blind, placebo-controlled phase 3 study The study is designed to compare the efficacy of stiripentol to a placebo in patients 6 years and older with primary hyperoxaluria type 1, 2 or 3.

The study will be conducted in 2 periods: a 6-month, placebo-controlled, double-blind treatment period (period 1) followed by a 6-month open-label treatment period with blind maintained on results (period 2).

Patients who benefit from the treatment after the first 12 months of study treatment will be proposed to enter the open-label extension (OLE) part of the study to continue to assess the long-term efficacy and safety of stiripentol.

ELIGIBILITY:
Screening Criteria :

* 1. Male or female patients aged ≥ 6 years at the time of consent signature
* 2. Diagnosed with primary hyperoxaluria (type 1, 2 or 3) documented as per standard methods
* 3. With last estimated Glomerular Filtration Rate ≥ 45 mL/min/1.73 m2
* 4. Able to understand and willing to comply with study requirements and to provide written informed consent. In case of patient under the age of legal consent, the legal guardian(s) must provide informed consent and the patient should provide assent as per local and national requirements
* 5. Female patients with contraception (intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, surgical sterilization of male partner, established use of oral, implantable, injectable, or transdermal hormonal methods of contraception, a double-barrier method (combination of male condom with cap, diaphragm, or sponge, in conjunction with spermicide) or true sexual abstinence

Inclusion Criteria:

* 1. Diagnosed with primary hyperoxaluria disease and subtype (type 1, 2 or 3) confirmed by genetic testing
* 2. Receiving optimal management of the disease through standard of care strategies (e.g., increased fluid intake, vitamin B6, potassium citrate) with or without approved target medications (e.g., lumasiran). Patients not receiving lumasiran can only be enrolled if they are not eligible for treatment with lumasiran for the specific following reasons: contraindications, previous treatment discontinued due to lack of efficacy or poor tolerability, not meeting national or regional eligibility criteria for treatment, investigator judgement
* 3. With mean 24-hour urinary oxalate excretion from 2 valid 24-hour urine collections ≥ 0.70 mmol/24h/1.73m²
* 4. With estimated Glomerular Filtration Rate ≥ 45 mL/min/1.73 m2 (Schwartz et al., 2009 in pediatric patients and CKD-EPI in adults)
* 5. Pubescent and adult female patients must have a negative urine or serum pregnancy test within 60 days prior to first dose of study treatment if of childbearing potential. If the urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible
* 6. In France, patient affiliated with or who benefits from a social security scheme

Exclusion Criteria:

* 1. Any relevant change in the use of any component of the standard of care (fluid intake, vitamin B6, potassium citrate) in the 4 weeks prior to inclusion or if such change is planned to occur during the first 6 months of the study
* 2. If under approved targeted medications (e.g., lumasiran), treatment should have been administered for at least 6 months, with no change in dose or regimen in the 3 months prior to inclusion or ifsuch change is planned it should not occur during the first 12 months of the study
* 3. History of kidney or liver transplant
* 4. Presenting any of the following liver function tests abnormalities during the screening period:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)> 2 × upper limit of normal (ULN)
  2. Total bilirubin > 1.5 x ULN. Patients with elevated total bilirubin that is secondary to documented Gilbert's syndrome are eligible if the total bilirubin is < 2 x ULN
* 5. Recent (4 weeks before the screening visit) or planned change in eating habits
* 6. Intermittent fasting planned during the 6 first months of the study period (e.g., Ramadan)
* 7. Other medical conditions or comorbidities, treatment, which in the opinion of the investigator, would interfere with study compliance or data interpretation
* 8. Presenting any significant biological or clinical anomalies that are not compatible with participation in the study according to the investigator
* 9. History of severe allergy, asthma, skin rashes, intolerance to lactose or hypersensitivity to the study treatments
* 10. Treatment affecting hepatic metabolism (i.e., cimetidine, ketoconazole, fluconazole, itraconazole, phenytoin, rifampicin, rifabutin) that is ongoing or has been taken in the month prior to the selection visit
* 11. Treatment affecting the renal tubule (probenecid, β-lactam, etc.,) that is ongoing or has been taken in the two weeks prior to the start of the study
* 12. Contraindications to stiripentol as defined in the applicable Investigator's Brochure (i.e. patients presenting a hypersensitivity to the active substance or any excipients)
* 13. Patient at risk of pregnancy, pregnant or breastfeeding female
* 14. Patient under guardianship or curatorship
* 15. Patient under the protection of the Court or deprived of liberty
* 16. Patient participating in another interventional clinical trial which could interfere with the trial's results or impact the other trial's results; or within the last 30 days or 5 half-lives of the study investigational treatment, whichever is longer, prior to the urinary sampling during the screening period, or are in follow-up of another clinical study prior to randomization
* 17. Patient whose current state of health does not allow him/her to give consent

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
% change in 24-hour urinary oxalate excretion corrected for body surface area (BSA) determined from 24-hour urine sample collections | % change in 24-hour urinary oxalate excretion between baseline value and value at month 6
  % change in 24-hour urinary oxalate excretion in mg/kg corrected for body surface area (BSA) between baseline and Month 6 and determined from 24-hour urine sample collections

SECONDARY OUTCOMES:
% change in 24-hour urinary oxalate excretion corrected for body surface area (BSA) determined from 24-hour urine sample collections | % change in 24-hour urinary oxalate excretion between baseline value and value at month 3
  % change in 24-hour urinary oxalate excretion in mg/kg corrected for body surface area (BSA) from baseline to Month 3 and determined from 24-hour urine sample collections
Absolute change in 24-hour urinary oxalate excretion in mg/kg corrected for body surface area (BSA) from baseline to Month 3 and Month 6 | Absolute change in 24-hour urinary oxalate excretion between baseline value to Month 3 and Month 6 values.
  Absolute change in 24-hour urinary oxalate excretion in mg/kg corrected for BSA from baseline to Month 3 and Month 6
Change in 24-hour urine oxalate/creatinine ratio from baseline to Month 3 and Month 6 | Change in 24-hour urine oxalate/creatinine ratio between baseline value to month 3 and month 6 values
  Concentration of 24-hour urine oxalate and 24-hour urine creatinine will be combined to report urine oxalate/creatinine ratio from baseline to Month 3 and Month 6. The concentrations will be determined using a validated assay
% of patients with urinary oxalate lower than 1.5 x upper limit of normal (ULN)) at Month 3 and Month 6 | At 3 and 6 months of treatment.
  %of patients with near normalisation of 24-hour urinary oxalate level corrected for BSA (defined as urinary oxalate lower than 1.5 x upper limit of normal (ULN)) at Month 3 and Month 6)
% of patients with normalisation of 24-hour urinary oxalate level corrected for bode surface area at Month 3 and Month 6 | At 3 and 6 months of treatment.
  % of patients with near normalisation of 24-hour urinary oxalate level corrected for BSA (defined as urinary oxalate lower than 1.5 x upper limit of normal (ULN)) at Month 3 and Month 6)
Blood samples for assessment of change in estimated glomerular filtration rate (eGFR in mL/min/1.73m2) from baseline to Month 6 | Change in estimated glomerular filtration rate (eGFR) between baseline value and month 6 value
  Blood samples for assessment of change in estimated glomerular filtration rate (eGFR). EGFR (mL/min/1.73m2) will be calculated from baseline to Month 6
Occurrence of and frequency of kidney stone events during the follow-up of the patient | From start of participation of the patient to end of the study (Month 60)
  Number of and frequency of kidney stone events reported during the follow-up of the patient
Change in urine oxalate/creatinine ratios as assessed in spot urine collections between baseline and Month 6 | From start of participation of the patient to end of the study (Month 60)
  Urine oxalate/creatinine ratios will be calculated from the oxalate and creatinine levels measured in spot urine collected during patients' hospitalizations or at home. The concentrations will be determined using a validated assay.
Change in biological parameters : oxalate concentration measured in urinary spots collections between baseline and Month 6 | From baseline to 6 months of treatment.
  Change in oxalate concentration, related to kidney stone formation, measured in urinary spots collections between baseline and Month 6
Change in biological parameters : creatinine concentration measured in urinary spots collections between baseline and Month 6 | From baseline to 6 months of treatment.
  Change in creatinine concentration, related to kidney stone formation, measured in urinary spots collections between baseline and Month 6
Absolute change in quality of life measured by the Pediatric Quality of Life Inventory (PedsQL) questionnaire | At baseline and every 6 months until the end of the study (Month 60)
  Absolute change in the Pediatric Quality of Life Inventory (PedsQL [the generic and kidney failure (KF) modules]) for patients < 18 years of age (at screening) which is a 23 items 5-point Likert scale from: 0 (Never) to 4 (Almost always). Scores are transformed on a scale from 0 to 100 so higher score means better health.
Absolute change in quality of life measured by the Kidney Disease Quality of Life Questionnaire (KDQOL) | At baseline and every 6 months until the end of the study (Month 60)
  Absolute changes in the Kidney Disease Quality of Life Questionnaire (KDQOL) for patients ≥ 18 years of age (at screening) which is a 36 items survey with five subscales. Scores are transformed on a scale from 0 to 100 so higher score means better health.
Change in quality of life measured by the Euro Quality of Life Health State Profile Questionnaire (EQ-5D) | At baseline and every 6 months until the end of the study (Month 60)
  Change in Euro Quality of Life Health State Profile Questionnaire (EQ-5D) is a standardized instrument consisting of a questionnaire. Scoring of the questionnaire is based on degrees of disability. Higher scores indicate better health status.
Change in quality of life measured by the Euro Quality of Life Health State Profile Visual Analog Scale (VAS) : EQ-5D | At baseline and every 6 months until the end of the study (Month 60)
  Change in EQ-5D Visual Analog Scale EQ-5D is a standardized instrument consisting of a visual analog scale pertaining to 5 dimensions. Scoring of the visual analog scale is based on a visual scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher scores indicate better health status.

OTHER OUTCOMES:
Height in meters | At baseline and every 3 months until the end of the study (Month 60)
  Changes in height in meters
Weight in kilograms | At baseline and every 3 months until the end of the study (Month 60)
  Changes in weight in kilograms
Changes in liver function tests (clinical laboratory parameters) | From start of participation of the patient to the end of the study
  Changes in liver function tests (AST, ALT, GGT, ALP, Bilirubin (total and direct))
Complete blood count with differential | At baseline and every months until the end of the study (Month 60)
  Changes in complete blood count with differential ( blood test results)
Frequency and nature of adverse events | From baseline to the end of the study (Month 60)
  Collect of the frequency and nature of adverse events
Change in 24-hour urinary glyoxylate, glycine and glycolate | From start of participation of the patient to end of the study (Month 60)
  Change in 24-hour urinary glyoxylate, glycine and glycolate
Change from baseline (percent and absolute) in 24-hour urine oxalate excretion, percentage of time that 24-hour urinary oxalate ≤ 1.5 x ULN, 24-hour urine oxalate/creatinine ratios and eGFR | From start of participation of the patient to end of the study (Month 60)
  Change from baseline (percent and absolute) in 24-hour urine oxalate excretion, percentage of time that 24-hour urinary oxalate ≤ 1.5 x ULN, 24-hour urine oxalate/creatinine ratios and eGFR
PK parameters : volume of distribution of stiripentol | From start of participation of the patient to end of the study (Month 60)
  PK parameters : volume of distribution of stiripentol based on appropriate PK sampling scheme (on Month 0, Month 6 and Month 12), and further determined through a population PK (popPK) approach
PK parameters : clearance of stiripentol | From start of participation of the patient to end of the study (Month 60)
  PK parameters : clearance of stiripentol based on appropriate PK sampling scheme (on Month 0, Month 6 and Month 12), and further determined through a population PK (popPK) approach
Exposure parameters : Peak Plasma Concentration (Cmax) of stiripentol | From start of participation of the patient to end of the study (Month 60)
  Peak Plasma Concentration (Cmax) of stiripentol based on appropriate PK sampling scheme (on Month 0, Month 6 and Month 12), and further determined through a population PK (popPK) approach
Exposure parameters : Minimum Plasma Concentration (Cmin) of stiripentol | From start of participation of the patient to end of the study (Month 60)
  Minimum Plasma Concentration (Cmin) of stiripentol based on appropriate PK sampling scheme (on Month 0, Month 6 and Month 12), and further determined through a population PK (popPK) approach
Exposure parameters : Area under the plasma concentration versus time curve (AUC) of stiripentol | From start of participation of the patient to end of the study (Month 60)
  Area under the plasma concentration versus time curve (AUC) of stiripentol based on appropriate PK sampling scheme (on Month 0, Month 6 and Month 12), and further determined through a population PK (popPK) approach
Change in plasma oxalate concentrations | At baseline and every three Months until month 12
  Change in plasma oxalate concentrations
Change in plasma vitamin B6 concentrations | At baseline and every three Months until month 12
  Change in plasma vitamin B6 concentrations
Change in nephrocalcinosis as assessed by kidney imaging | At baseline and every 6 months until the end of the study (Month 60)
  Change in nephrocalcinosis as assessed by kidney imaging
Change in bone conditions during the follow-up | At Baseline and at Month 3,6 and 12
  Change in bone conditions during the follow-up based on questions from the investigator to the patient collected in the CRF
Prediction of urinary oxalate excretion at exposure of clinical interest for stiripentol from a PK/PD model | At baseline and every 6 months until month 12
  Prediction of urinary oxalate excretion at exposure of clinical interest for stiripentol from a PK/PD model
Change in patient, caregiver and investigator impact and experiences as evaluated by patient and investigator experience surveys | At baseline and every 6 months until end of the study (Month 60)
  Change in patient, caregiver and investigator impact and experiences as evaluated by patient and investigator experience surveys

CONTACTS AND LOCATIONS:
Overall Officials: Oana BERNARD, MD, Study Director — Chief Scientific Officer